CLINICAL TRIAL: NCT03660800
Title: An Open-label, Single-Dose, Safety, Tolerability and Pharmacokinetic Study of Oral CTAP101 (Calcifediol) Extended-release Capsules in Japanese and Non-Japanese Healthy Subjects
Brief Title: Pharmacokinetics and Safety Study of CTAP101 Capsules in Japanese and Non-Japanese Healthy Subjects and Non-Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTAP101-CL-1020
Record Dates: First submitted 2018-08-23; First posted 2018-09-07 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Vitamin D Insufficiency; Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CTAP101 Capsules 450mcg/weekly fasted (Experimental)
  Interventions: Drug: CTAP101 Capsules
- CTAP101 Capsules 900mcg/weekly fasted (Experimental)
  Interventions: Drug: CTAP101 Capsules
- CTAP101 Capsules 1800mcg/weekly fasted (Experimental)
  Interventions: Drug: CTAP101 Capsules
- CTAP101 Capsules 900mcg/weekly fed (Experimental)
  Interventions: Drug: CTAP101 Capsules

INTERVENTIONS:
Drug: CTAP101 Capsules — Calcifediol Extended-Release Capsules

SUMMARY:
Pharmacokinetics and Safety Study of CTAP101 Capsules in Japanese and non-Japanese Healthy Subjects

DETAILED DESCRIPTION:
An Open-label, Single-Dose, Safety, Tolerability and Pharmacokinetic Study of Oral CTAP101 (Calcifediol) Extended-release Capsules in Japanese and non-Japanese Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Signed the informed consent form as described in Appendix 3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
2. Willing and able to comply with study instructions and to commit to all study days
3. Man or woman, 18 to 55 years of age inclusive at the time of signing the informed consent form
4. Overtly healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests
5. Body mass index (BMI) within 18.0 to 30.0 kg/m2 (inclusive) and body weight not less than 50 kg
6. Blood pressure (after at least 2 minutes of rest) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic.
7. A 12-lead ECG consistent with normal cardiac conduction and function, including:

   * Sinus rhythm
   * Pulse rate between 40 and 100 beats per minute (bpm)
   * QTc interval ≤450 milliseconds (QT interval corrected using Fridericia correction method [QTcF]
   * QRS interval of <120 milliseconds
   * PR interval <200 milliseconds
   * Morphology consistent with healthy cardiac conduction and function
8. Must have negative tests for drugs of abuse at Screening and Day -2
9. Must have a negative alcohol test at Screening and Day -2
10. Must have adequate venous access in both arms, in the opinion of the Investigator
11. Has a screening serum total 25-hydroxyvitamin D level between 10 and 40 ng/mL, inclusive
12. If male, must agree to use contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period
13. If female, be sterile (ie, at least 1 month post-surgical sterilization, confirmed nonsurgical sterilization or at least 6 months post-menopausal [as determined by follicle stimulating hormone (FSH) / estradiol testing]); or who are of childbearing potential but are abstinent, have a surgically sterile partner (ie, at least 6 months postvasectomy), or are using a copper intrauterine device or a combination of at least 2 acceptable barrier methods such as condom + intravaginal spermicide, diaphragm + intravaginal spermicide, or cervical cap + intravaginal spermicide. Contraceptive medications (oral or by other routes) containing steroid hormones are not allowed. Women of childbearing potential must not be lactating and must have a negative pregnancy test at screening and Day -2, and agree to continue their accepted method of contraception throughout the study. See guidance on contraceptives in Appendix 5. Additional Inclusion Criteria for Japanese Participants Only

1. Be first generation Japanese defined as:

* Born in Japan
* Has 2 Japanese biological parents and 4 Japanese biological grandparents
* Has lived outside of Japan for less than 5 years
* Has made no significant changes in lifestyle, including diet, since leaving Japan Additional Inclusion Criteria for non-Japanese Participants Only

  1. Not of Japanese or Asian descent
  2. Parents and grandparents not born in Japan or in any Asian countries Note: Retesting of abnormal lab values that may lead to exclusion will be allowed once.

Retesting will take place during an unscheduled visit during the screening phase.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has taken a Vitamin D supplement within 28 days prior to dosing
2. Has a medically confirmed history of kidney stones within the previous 2 years
3. Has a urine calcium: creatinine ratio > 0.2 at the Screening visit
4. Has a known or suspected hypersensitivity to any of the constituents of the investigational products
5. Has a history of or current clinically significant medical illness including but not limited to, cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); lipid abnormalities; significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; hepatic or renal insufficiency (creatinine clearance below 60 mL/min); thyroid disease; neurologic or psychiatric disease; infection; or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results.
6. Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening as deemed appropriate by the investigator
7. Clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening as deemed appropriate by the investigator
8. Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
9. Has received an investigational drug or used an invasive investigational medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before Day 1.
10. Has donated 1 unit (450 mL) or more of blood or plasma within 30 days of dosing
11. Has an acute illness within 5 days prior to the first dose of study medication
12. Has received any prescribed systemic or topical medication within 14 days of dosing, received a vaccination within 30 days of dosing, or taken any nonprescription systemic or topical medication or herbal preparation within 7 days of dosing (exception: occasional use of acetaminophen or ibuprofen at nonprescription doses).
13. History of drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) criteria within 5 years before Screening or positive test result(s) for alcohol and/or drugs of abuse (including prescription drugs such as stimulants, opioids, and benzodiazepines) at Screening or at Admission on Day -2
14. Has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level >1.5 times the upper limit of normal (ULN), active liver disease or jaundice at Screening or Day -2
15. Is considering or has preplanned surgery or procedures that would interfere with the conduct of the study
16. Is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related AEs as assessed by industry standards | 8 weeks
  Incidence of AEs will be summarized by arm for all treatment-emergent AEs. Number and percent of participants with AEs will be summarized by system organ class and preferred term and presented overall and by arm.
Change in baseline of peak plasma concentration | 8 weeks
  Baseline finding will be measured against the different time points collected
Change in mean total of the different components of calcifediol | 8 weeks
  Descriptive statistics will be calculated for PD assessment in the per protocol population.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Mussallem, Study Chair — WCCT Global, Inc
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No